CLINICAL TRIAL: NCT01413542
Title: Pharmacogenetics of Ace Inhibitor-Associated Angioedema:Aim 1
Brief Title: Pharmacogenetics of Ace Inhibitor-Associated Angioedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Chair of Dept of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HL079184; NCT00139503 (obsolete NCT alias)
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Results first posted 2015-11-04 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension; Diabetes Type 2
Keywords: DPPIV inhibitors; ACE inhibitors; Bradykinin; glucagon-like peptide (GLP-1); BNP; diabetes; hypertension
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; Substance P; Bradykinin; Enalaprilat; Angiotensin-Converting Enzyme Inhibitors; Glucagon-Like Peptide 1; Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo then sitagliptin (DPP4 inhibition) group 1 (Placebo Comparator): The effect of vehicle and enalaprilat on the forearm blood flow and t-PA responses to bradykinin and substance P are studied after administration of placebo or sitagliptin (DPP4 inhibition).
  Interventions: Drug: Sitagliptin (DPP4 inhibitor); Drug: Substance P,; Drug: bradykinin; Drug: enalaprilat (ACE inhibitor)
- Sitagliptin (DPP4 inhibition) then placebo group 1 (Placebo Comparator): The effect of vehicle and enalaprilat (ACE inhibition) on the forearm blood flow and t-PA responses to substance P and bradykinin are studied after administration of sitagliptin (DPP4 inhibition) or placebo
  Interventions: Drug: Sitagliptin (DPP4 inhibitor); Drug: Substance P,; Drug: bradykinin; Drug: enalaprilat (ACE inhibitor)
- Placebo then sitagliptin group 2 (Placebo Comparator): The effect of vehicle and enalaprilat (ACE inhibition) on the forearm blood flow and t-PA responses to glucagon-like peptide-1 and brain natriuretic pepdie are studied after administration of placebo or sitagliptin (DPP4 inhibition).
  Interventions: Drug: Sitagliptin (DPP4 inhibitor); Drug: Glucagon-like peptide 1; Drug: brain natriuretic peptide
- Sitagliptin (DPP4 inhibition) then comparator group 2 (Placebo Comparator): The effect of vehicle and enalaprilat on the forearm blood flow and t-PA responses to glucagon-like peptide and brain natriuretic peptide are studied after administration of placebo or sitagliptin (DPP4 inhibition).
  Interventions: Drug: Sitagliptin (DPP4 inhibitor); Drug: Glucagon-like peptide 1; Drug: brain natriuretic peptide

INTERVENTIONS:
Drug: Sitagliptin (DPP4 inhibitor) — Sitagliptin 200 mg (DPP4 inhibitor) or matching placebo will be given one hour prior to intra-arterial infusions
  Other Names: Januvia
Drug: Substance P, — Substance P intra-brachial artery (2,4,8 pmol/min)
  Arms: Placebo then sitagliptin (DPP4 inhibition) group 1; Sitagliptin (DPP4 inhibition) then placebo group 1
Drug: bradykinin — bradykinin intra-brachial artery (23.6, 47.2, and 94.3 pmol/min)
  Arms: Placebo then sitagliptin (DPP4 inhibition) group 1; Sitagliptin (DPP4 inhibition) then placebo group 1
Drug: enalaprilat (ACE inhibitor) — intra-brachial artery(0.33 µg/min per 100 mL forearm volume)
  Other Names: vasotec
  Arms: Placebo then sitagliptin (DPP4 inhibition) group 1; Sitagliptin (DPP4 inhibition) then placebo group 1
Drug: Glucagon-like peptide 1 — intra-brachial artery (0.45-3.60 pmol/min)
  Other Names: GLP-1
  Arms: Placebo then sitagliptin group 2; Sitagliptin (DPP4 inhibition) then comparator group 2
Drug: brain natriuretic peptide — Intra-brachial artery (0.90, 1.80 and 3.6 pmol/min)
  Other Names: nesiritide
  Arms: Placebo then sitagliptin group 2; Sitagliptin (DPP4 inhibition) then comparator group 2

SUMMARY:
The investigators would like to find out if sitagliptin (dipeptidyl peptidase-4 or DPP4 inhibition), a drug to treat diabetes, affects blood vessel relaxation in healthy people receiving enalapril (angiotensin converting enzyme or ACE inhibition), a blood pressure medicine. Understanding how these drugs interact in healthy people will help us learn their potential effects in people who have diabetes.

DETAILED DESCRIPTION:
To test the hypothesis that DPPIV inhibition with sitagliptin potentiates the vasodilator response to substance P in the presence of ACE inhibition with enalaprilat and to BNP and GLP-1 even in the presence of ACE inhibition. The aim promises to provide important new data regarding the mechanism of action of DPPIV inhibitors and interactive effects of these two drug classes used in a growing population of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 inclusive
* Men and women
* Black and White Americans
* BMI <25

For female subjects:

* Postmenopausal status for at least 1 year
* Status post surgical sterilization
* If childbearing potential, utilization of a barrier method of birth control and willingness to undergo blood B-hcg testing prior to drug treatment and on every study day

Exclusion Criteria:

* Smoking
* Diabetes type 1 or 2, as defined by a fasting glucose of 126 mg/dl or greater or the use of anti-diabetic medication
* Hypertension as defined by an untreated seated SBP greater than 140 mmHg an untreated DBP greater than 90 mmHg or the use of antihypertensives
* History of reported or recorded hypoglycemia (plasma glucose less than 70 mg/dl)
* Pregnancy
* Breast-feeding
* Use of hormone replacement therapy
* The use of contraceptive therapy
* Use of any medication other than multivitamin
* Hematocrit <35%
* Cardiovascular disease such as history of myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure(LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
* Asthma
* History of angioedema
* History of cough or other side effect during ACE inhibitor use
* Impaired renal function, as defined by an eGFR<60ml/min/1.73M2
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Impaired hepatic function (aspartate amino transaminase[AST] and/or alanine amino transferase [ALT]>2 x upper limit of normal range
* History of alcohol or drug abuse
* Treatment with any investigational drug in the 1 month preceding the study
* Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return to follow-up visits, and the unlikelihood of completing the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University- General Clinic Research Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Devin JK, Pretorius M, Nian H, Yu C, Billings FT 4th, Brown NJ. Dipeptidyl-peptidase 4 inhibition and the vascular effects of glucagon-like peptide-1 and brain natriuretic peptide in the human forearm. J Am Heart Assoc. 2014 Aug 26;3(4):e001075. doi: 10.1161/JAHA.114.001075. PMID 25158865
- [Derived] Devin JK, Pretorius M, Nian H, Yu C, Billings FT 4th, Brown NJ. Substance P increases sympathetic activity during combined angiotensin-converting enzyme and dipeptidyl peptidase-4 inhibition. Hypertension. 2014 May;63(5):951-7. doi: 10.1161/HYPERTENSIONAHA.113.02767. Epub 2014 Feb 10. PMID 24516103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 participants were enrolled in this study (23 in Group 1 and 21 in Group 2) and completed screening procedures. Twelve of 23 participants met inclusion and exclusion criteria and completed all study-related procedures in Group 1. Seventeen of 21 participants met inclusion/exclusion criteria and completed all study-related procedures in Group 2.
Groups:
- Placebo Then Sitagliptin (DPP4 Inhibibition)=Group 1: Participants first received Placebo then Sitagliptin 200 mg by mouth one time on each of two study days. Two weeks separated each study day. Each study day examined the effect of vehicle and enalaprilat on the forearm blood flow and tPA responses to bradykinin and substance P.
- Sitagliptin (DPP4 Inhibition) Then Placebo=Group 1: Participants first received Sitagliptin 200 mg then Placebo by mouth one time on each of two study days. Two weeks separated each study day. Each study day examined the effect of vehicle and enalaprilat on the forearm blood flow and tPA responses to bradykinin and substance P.
- Placebo Then Sitagliptin (DPP4 Inhibition)=Group 2: Participants first received Placebo then Sitagliptin 200 mg by mouth one time on each of two study days. Two weeks separated each study day. Each study day examined the forearm blood flow and tPA responses to brain natriuretic peptide (BNP) and glucagon-like receptor 1 (GLP-1).
- Sitagliptin (DPP4 Inhibition) Then Placebo = Group 2: Participants first received Sitagliptin 200 mg then Placebo by mouth one time on each of two study days. Two weeks separated each study day. Each study day examined the forearm blood flow and tPA responses to brain natriuretic peptide (BNP) and glucagon-like receptor 1 (GLP-1).
Period: Overall Study
Arm/Group | Placebo Then Sitagliptin (DPP4 Inhibibition)=Group 1 | Sitagliptin (DPP4 Inhibition) Then Placebo=Group 1 | Placebo Then Sitagliptin (DPP4 Inhibition)=Group 2 | Sitagliptin (DPP4 Inhibition) Then Placebo = Group 2
Started | 6 | 6 | 9 | 8
Completed | 5 | 6 | 6 | 7
Not Completed | 1 | 0 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This population represents the 29 participants (12 in Group 1; 17 in Group 2) who passed screening and completed at least one study arm. 1 subject did not complete the 2nd arm in Group 1. 4 subjects did not complete the second arm in Group 2. Results and baseline characteristics are presented inclusive of these patients.
Groups:
- Group 1: Participants were randomized to sitagliptin 200 mg vs. placebo on each of two study days. On each study day, the effects of vehicle and enalaprilat on forearm blood flow and tPA responses to bradykinin and substance P were studied.
- Group 2: Participants were randomized to sitagliptin 200 mg vs. placebo on each of two study days. On each study day, the effect of brain natriuretic peptide and glucagon like receptor-1 (GLP-1) on forearm blood flow and tPA release was studied.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12.0) | 35.4 (10.0) | 36.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 9 | 12 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: The Effect of Enalaprilat (ACE Inhibition), Sitagliptin (DPP4 Inhibition), or the Combination on the Vasodilator Response (Forearm Blood Flow) to Substance P (SP) and Bradykinin (Group 1) or Glucagon Like Peptide-1 and Brain Naturetic Peptide (Group 2).
Description: Forearm blood flow (FBF) was measured by strain gauge plethysmography at the completion of each dose of intra-arterial peptide. A dose response curve was therefore constructed for each vasoactive peptide substrate. The effect of sitagliptin (DPP4 inhibition) vs. placebo and enalaprilat (ACE inhibition) vs. vehicle on the forearm blood flow response to each peptide could then be determined.
Time Frame: 60 minutes post-placebo or sitagliptin (DPP4 inhibition) and over last 2 minutes of each 5 min infusion per peptide dose (30 min washout between peptides); sequence repeated with enalaprilat (ACE inhibition) or vehicle
Population: In Group 1: Peptide 1=Max dose Bradykinin; Peptide 2=Substance P (SP) In Group 2: Peptide 1=GLP-1; Peptide 2=BNP (FBF expressed as percent change for both peptides) ACE inhibition=enalaprilat DPP4 inhibition=sitagliptin
Measure: Mean (95% Confidence Interval); unit: estimate of difference(ml/min/100ml FBF)
Groups:
- Group 1: Participants were randomized to sitagliptin 200 mg (DPP4 inhibitor) vs. placebo on each of two study days. On each study day, the effects of vehicle and enalaprilat (ACE inhibitor) on forearm blood flow and tPA responses to bradykinin (peptide 1) and substance P (SP) (peptide 2) were studied.
- Group 2: Participants were randomized to sitagliptin 200 mg (DPP4 inhibitor) vs. placebo on each of two study days. On each study day, the effect of study drug on FBF response to glucagon like peptide-1 (peptide 1) and brain natriuretic peptide (peptide 2) was studied.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 12 | 17
estimate of difference(ml/min/100ml FBF)
  Effect ACE inhibition on FBF response to Peptide 1 | 6.5 [4.0 to 9.0] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 1 is not a substrate of ace
  Effect DPP4 inhibition on FBF Response to Peptide1 | 0.2 [-2.4 to 2.7] | -5.0 [-11.6 to 1.6]
  Effect ACE/DPP4 inhibit on FBF response Peptide 1 | 5.9 [3.3 to 8.4] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 1 is not a substrate of ace
  Effect DPP4/ACEinhib vs. ACEinhib (FBF to Pep1) | -0.6 [-3.1 to 1.9] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 1 is not a substrate of ace
  Effect DPP4/ACEinhib vs. DPP4inhib (FBF to Pep1) | 5.7 [3.2 to 8.2] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 1 is not a substrate of ace
  Effect ACE inhibition on FBF response to Peptide 2 | 0.8 [-0.3 to 2.0] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 2 is not a substrate of ace
  Effect DPP4 inhibition on FBF response to Peptide2 | 0.1 [-0.1 to 1.3] | -3.2 [-37.4 to 31.0]
  Effect ACE/DPP4 inhibition on Peptide 2 FBF | 0.6 [-0.6 to 1.7] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 2 is not a substrate of ace
  Effect DPP4/ACEinhib vs. ACEinhib (FBF to Pep2) | -0.3 [-1.4 to 0.9] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 2 is not a substrate of ace
  Effect DPP4/ACEinhib vs. DPP4inhib (FBF to Pep2) | 0.4 [-0.8 to 1.6] | NA [NA to NA] — effect of ace inhibition not studied in this group as peptide 2 is not a substrate of ace
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Group 1: The effect of treatment (placebo, ACE or DPP4 inhibitor, or the combination) on vasodilator response to peptide, measured as forearm blood flow was determined. Group 2: The effect of treatment (placebo, DPP4 inhibitor) on vasodilator response to peptide, measured as percent change in forearm blood flow was determined; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Effect of ACE inhibition on FBF response to bradykinin (p<0.001). Other comparisons: Effect of DPP4 inhibition on FBF response to bradykinin (p=0.89); Effect of ACE (p=0.16), DPP4 (p=0.82), or combined inhibition (p=0.35) on FBF response to sub P; Effect of DPP4 inhibition on vasodilator response to GLP-1 (p=0.14) or BNP (p=0.85). p<0.05 threshold for statistical significance; Estimate of Difference

2. Secondary Outcome: Assess Tissue Type Plasminogen Activator (tPA) Release
Description: Following measurement of FBF, samples will be obtained to determine the effect of ACE inhibition and/or DPP4 inhibition on tPA release in response to bradykinin and substance P (SP) (group 1)
Time Frame: Blood for analysis of tPA release was obtained 60 minutes after sitagliptin (DPP4 inhibition) vs. placebo and after each assessment of FBF (see primary outcome measure)
Measure: Number (95% Confidence Interval); unit: estimate of difference (ng/min/100mL)
Groups:
- Group 1 (Males); Group 1 (Females): The effect of ACE inhibition and/or DPP4 inhibition on tPA release in response to bradykinin and substance P (SP) was evaluated.
Arm/Group | Group 1 (Males) | Group 1 (Females)
Number analyzed (Participants) | 5 | 7
estimate of difference (ng/min/100mL)
  Effect ACE inhibition on bradykinin tPA release | 118.6 [78.9 to 158.4] | 145.5 [107.0 to 184.1]
  Effect of DPP4 inhibition on bradykinintPA release | 1.6 [-38.6 to 41.8] | 12.9 [-26.5 to 52.3]
  Effect of ACE/DPP4 inhibitio on bradykinin tPA | 90.9 [50.8 to 131.0] | 132.1 [93.8 to 170.5]
  effect ace/dpp4 vs. aceinhibi on bradykinin tpa | -27.8 [-68.2 to 12.6] | -13.4 [-52.1 to 25.3]
  effect ace/dpp4 vs. dpp4inhib on bradykinin tpa | 89.3 [48.5 to 130.1] | 119.3 [80.2 to 158.3]
  Effect of ACE inhibition on SP tPA release | -15.3 [-41.8 to 11.3] | 43.9 [19.8 to 68.1]
  Effect of DPP4 inhibition on SP tPA | -25.8 [-52.4 to 0.8] | -29.0 [-53.4 to -4.6]
  Effect of ACE+DPP4 inhibition on SP tPA | 0.8 [-25.8 to 27.3] | 3.8 [-20.5 to 28.2]
  effect ace/dpp4 vs. aceinhibi on SP tpa | 16.1 [-10.5 to 42.6] | -40.1 [-64.5 to -15.7]
  effect ace/dpp4 vs. dpp4inhibi on SP tpa | 26.6 [0.0 to 53.1] | 32.8 [8.6 to 57.1]
Statistical Analysis 1: Comparison: Group 1 (Males) vs Group 1 (Females); Test type: Superiority or Other; p = 0.02, Mixed Models Analysis — Effect of DPP4 inhibition on tPA release during sub P in women (p=0.02 vs. placebo).Effect of ACE inhibition on tPA release during sub P in women (p<0.001); effect of DPP4 inhibition on tPA release during sub P and (p=0.001 vs. ACE inhibition alone); p<0.05 threshold for statistical significance

3. Secondary Outcome: Assess Effect of ACE and/or DPP4 Inhibition on Heart Rate Response to Substance P (SP)
Time Frame: Heart rate was measured every 5 minutes throughout the study day (and thus during each dose of peptide infusion)
Measure: Mean (Standard Error); unit: beats per minute
Groups:
- Group 1: The effect of ACE and/or DPP4 inhibition on change in heart rate in response to substance P (SP) was evaluated.
Arm/Group | Group 1
Number analyzed (Participants) | 12
beats per minute
  Change in Pulse after SP during Placebo | -1.8 (1.76)
  Change in Pulse after SP w/ACE inhibition | 2.55 (1.04)
  Change in Pulse after SP w/DPP4inhibition | 0.45 (1.74)
  Pulse change after SP w/ACE+DPP4inhibition | 4.55 (1.87)
Statistical Analysis 1: Comparison: Group 1; Test type: Superiority or Other; p = 0.011, Wilcoxon signed rank — Effect of combined ACE and DPP4 inhibition on change in heart rate in response to max dose substance P (p=0.011 vs placebo; ); p<0.05 threshold for statistical significance

4. Secondary Outcome: Effect of Treatment (ACE or DPP4 Inhibition, or Combined) on Norepinephrine (NE) Release (Arterial Venous Gradient) in Response to Substance P (SP)
Time Frame: Blood for analysis of norepinephrine (NE) release was obtained 60 minutes after sitagliptin (DPP4 inhibition) vs. placebo and after each assessment of FBF (see primary outcome measure)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Group 1
Number analyzed (Participants) | 12
pg/mL
  Change NE AV Gradient with SP after placebo | -43.18 (8.95)
  Change NE AV Gradient with SP after ACEinhibition | -52.18 (18.34)
  Change NE AV Gradient with SP after DPP4inhibition | -37.27 (12.21)
  Change NE AV with SP after ACE+DPPinhibition | 23.45 (31.47)
Statistical Analysis 1: Comparison: Group 1; Test type: Superiority or Other; p = 0.05, Wilcoxon signed rank — Effect of combined DPP4 and ACE inhibition on the change in the norepinephrine AV gradient during substance P as compared to treatment with placebo
Statistical Analysis 2: Comparison: Group 1; Test type: Superiority or Other; p = 0.007, Wilcoxon signed rank — Effect of combined DPP4 and ACE inhibition on the change in the norepinephrine AV gradient during substance P as compared to treatment with ACE inhibition alone (p=0.007)

5. Secondary Outcome: Effect of Treatment (DPP4 Inhibition vs. Placebo) on Venous GLP-1 Levels in Response to Arterial GLP-1 Infusion
Time Frame: Blood for analysis of GLP-1 levels was obtained one hour after sitagliptin (DPP4 inhibition) vs. placebo administration and after each dose of GLP-1
Measure: Mean (Standard Error); unit: pmol/L
Groups:
- Group 2: The effect of treatment (placebo vs. DPP4 inhibition) on venous GLP-1 levels during intra-arterial GLP-1 infusion.
Arm/Group | Group 2
Number analyzed (Participants) | 14
pmol/L
  Venous GLP-1 levels 1 hour after placebo | 5.13 (1.05)
  Venous GLP-1 Levels after Max Dose GLP-1 (Placebo) | 15.44 (2.94)
  Venous GLP-1 levels 1 hour after DPP4 inhibition | 5.39 (0.99)
  Venous GLP-1 levels Max Dose GLP-1 (DPP4inhibiton) | 30.63 (3.40)
Statistical Analysis 1: Comparison: Group 2; Test type: Superiority or Other; p = 0.01, wilxocon signed rank test — Effect of intra-arterial GLP-1 on venous GLP-1 concentrations during placebo (p=0.01)
Statistical Analysis 2: Comparison: Group 2; Test type: Superiority or Other; p = 0.01, Wilcoxon signed rank — Effect of intra-arterial GLP-1 on venous GLP-1 concentrations during sitagliptin (p=0.01)
Statistical Analysis 3: Comparison: Group 2; Test type: Superiority or Other; p = 0.04, Wilcoxon signed rank — Effect of DPP4 inhibition on venous GLP-1 levels at high dose of intra-arterial GLP-1 (p=0.04 vs. placebo)

ADVERSE EVENTS:
Description: 1 Subject (Group 1) did not complete sitagliptin arm due to inability to establish arterial access.
  1 Subject (Group 2) did not complete placebo arm because the Investigator withdrew them after Serious Adverse Event.
  3 Subjects (Group 2) did not complete the sitagliptin arm due to inability to establish arterial access during the sitagliptin arm.
Groups:
- Group 1 (Placebo Arm); Group 1 (Sitagliptin Arm): Participants were randomized to sitagliptin 200 mg vs. placebo on each of two study days. On each study day, the effects of vehicle and enalaprilat on forearm blood flow and tPA responses to bradykinin and substance P were studied.
- Group 2 (Placebo Arm); Group 2 (Sitagliptin Arm): Participants were randomized to sitagliptin 200 mg vs. placebo on each of two study days. On each study day, the effect of brain natriuretic peptide and glucagon like receptor-1 (GLP-1) on forearm blood flow and tPA release was studied.
Arm/Group | Group 1 (Placebo Arm) | Group 1 (Sitagliptin Arm) | Group 2 (Placebo Arm) | Group 2 (Sitagliptin Arm)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/16 | 1/14
Other Adverse Events (participants affected / at risk) | 3/12 | 2/11 | 3/16 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Placebo Arm) (N=12) | Group 1 (Sitagliptin Arm) (N=11) | Group 2 (Placebo Arm) (N=16) | Group 2 (Sitagliptin Arm) (N=14)
Orthostasis with Syncopal Event (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Placebo Arm) (N=12) | Group 1 (Sitagliptin Arm) (N=11) | Group 2 (Placebo Arm) (N=16) | Group 2 (Sitagliptin Arm) (N=14)
Swelling of instrumented arm (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — One woman experienced angioedema of the instrumented forearm after infusion of bradykinin and substance P on the sitagliptin treatment day.
Transient Lightheadedness (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Within 2 weeks of completion of first study day.
Neuropraxia in the instrumented arm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Resolved over 2 weeks without therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No